CLINICAL TRIAL: NCT04679181
Title: Acceptability Assessment of an "Organization of Care Integrating Artificial Intelligence and a Solution of Telemedicine" on Care of the Nursing Home Residents Located in a Medical Desert: Pilot Study INTEL@MED-POC
Acronym: Intel@Med-Poc
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 87RI18-0018/Intel@Med-Poc
Record Dates: First submitted 2020-12-03; First posted 2020-12-22 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-04

CONDITIONS: Homes for the Aged
Keywords: aged; telemedicine; artificial intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active arm (Experimental): use of telemedicine
  Interventions: Other: Telemedecine

INTERVENTIONS:
Other: Telemedecine — telemedical consultation

SUMMARY:
While depend elderly people needs are important in Nursing Home, the medical resources are weak from both inside and outside residences located in a medical desert. The goal of this project is to measure the acceptability of Artificial Intelligence and Telemedicine in Nursing Home located in medical desert for patients, nurses, and medical doctor

DETAILED DESCRIPTION:
The ageing of the population comes along with the problematic of chronic pathologies and dependence, with sometimes serious consequences resulting in an admission in Nursing Home. While the low require a medical doctor in each Nursing Home, one third of the Nursing Home does not have. Some Nursing Homes can be in a tricky situation with no medical doctor coordinator and the difficulty of access to a medical doctor who covered a wide territory. In this context, the emergence of Artificial Intelligence coupled with Telemedicine is a new opportunity to find solution in healthcare organization and to develop advanced geriatric medical practice in medical desert territory. The goal of this study is to quantify and characterize the acceptability of Artificial Intelligence and Telemedicine in Nursing Home located in medical desert for patients, nurses, and medical doctor.

All the patients were examined by a nurse. The symptoms filled by the nurse in the Artificial Intelligence/Telemedicine device are sent and then analyzed by a distant medical doctor to purpose a care. The nurse also solicited the attending medical doctor as usual care.

The recommendations of the both medical doctors could be (i) Vital emergency, (ii) non-vital emergency necessitate medication or hospitalization, and (iii) non-emergency with medical appointment.

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 65 years old.
* Patient living in Nursing Home located in medical desert.
* Patient presenting symptoms involved medical doctor call.
* Patient or legal representative having signed consent form
* Patient covered by social security

Exclusion Criteria:

* End of life patient.
* Chronic aphasic patient.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2023-03-25 (Estimated); Study Completion 2023-03-25 (Estimated)

PRIMARY OUTCOMES:
Acceptability for nurse to use Artificial Intelligence / Telemedecine device analyzed by distant medical doctor | 13 months
  Proportion of the Artificial Intelligence / Telemedecine utilization by the nurse vs medical doctor as usual care
Number of non-programmed hospitalization for both distant medical doctor and usual care recommendations | 13 months
  Comparison of non programmed hospitalization in both distant medical doctor analysis and medical doctor as usual care
delay to obtain the medical expertise | 13 months
  Comparison of time to obtain the medical expertise for distant medical doctor and usual care recommandations

SECONDARY OUTCOMES:
sensitivity and specificity of diagnostic | 13 months
  Calculation of sensitivity and specificity of diagnostic for acute disease and emergency for both distant medical doctor and usual care recommendations

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - EHPAD Le Bois Joli, Auzances
  - EHPAD Le Chant des Rivières, Chambon-sur-Voueize
  - EHPAD La Porte d'Aquitaine, La Roche-Chalais
  - Ehpad Le Chavanon, Merlines
  - EHPAD Ernest Coulaud, Peyrelevade
  - EHPAD J et M Colaud, Saint-Privat

IPD SHARING:
Plan to Share IPD: No